CLINICAL TRIAL: NCT02983916
Title: Laparoscopic Adhesiolysis for Chronic Abdominal Pain Revisited
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RU-RTB-0005
Record Dates: First submitted 2016-11-23; First posted 2016-12-06 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2016-11

CONDITIONS: Chronic Pain; Tissue Adhesion
Keywords: Adhesions; Adhesiolysis; chronic pain; post-operative complications; anti-adhesion barrier; cine-MRI; shared decision making
MeSH Terms: conditions — Chronic Pain; Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: adhesiolysis: Group 1 (the operative group) consisted of all patients who underwent laparoscopy and/or laparotomy. Typically patients had positive cine-MRI. A few patients with inconclusive cine-MRI who underwent diagnostic laparoscopy are also included in this group. Patients with no adhesions found during operation remain in group 1, because analysis is performed on intention-to-treat basis.
  Interventions: Procedure: Adhesiolysis
- Group 2: Adhesions, conservative: Patients with evidence of adhesions based on cine-MRI who did not undergo laparoscopy or laparotomy.
- Group 3: No adhesions: Patients in whom no evidence of adhesions was found on cine-MRI, and who did not undergo laparoscopy or laparotomy .

INTERVENTIONS:
Procedure: Adhesiolysis — Diagnostic laparoscopy or laparotomy with lysis of adhesions.
  Groups: Group 1: adhesiolysis

SUMMARY:
Chronic abdominal and pelvic pain is a common complaint following peritoneal surgery, affecting 20-40% of patients. Adhesions account for 60% of chronic postoperative pain cases, suggesting that adhesiolysis can play an important role in the management of such pain. Despite initial promising results regarding the effect of adhesiolysis on post-operative pain, implementation of the procedure has been challenging. The major problems associated with adhesiolysis for pain are recurrence of pain, need for invasive diagnosis with high rates of 'negative' laparoscopies, and inadvertent bowel injury during surgery. However, diagnosis and treatment of adhesions may be improved through the use of novel cine-MRI techniques, and with application of anti-adhesion barriers following adhesiolysis.

In this study the investigators evaluate a new practice-based approach to the problem of chronic post-operative pain caused by adhesions. This practice-based approach includes use of a novel imaging technique for adhesions (cine-MRI) and shared decision making. Cine-MRI holds promise to diagnose and map adhesions. Thus patients with no adhesions, or high risk for bowel injury, can be waived from surgical treatment. By using anti-adhesion barriers the investigators attempt to prevent adhesion reformation and improve long-term outcomes of adhesiolysis.

DETAILED DESCRIPTION:
Laparoscopic adhesiolysis for chronic abdominal pain revisited.

Background Prevalence of chronic pain following abdominal surgery may be as high as 40%. Postoperative chronic pain can be caused by various reasons, but adhesions are identified as the most likely cause in more 60% of cases. Early studies of adhesiolysis reported high success rates, up to 80%, in patients with no other cause of pain. Nonetheless, adhesiolysis is now seldom used in the treatment of chronic abdominal pain. Controversy over laparoscopic adhesiolysis as treatment for abdominal pain was raised by the landmark trial of Swank et al. In this trial 100 patients were randomized after the diagnosis of adhesions was confirmed laparoscopy between adhesiolysis or diagnostic laparoscopy alone. In the adhesiolysis group 57% of patients reported long-term pain relief vs. 42% in the diagnostic group; this difference was not statistically significant. The authors concluded that adhesiolysis was not effective, and thereafter many surgeons discarded adhesiolysis as treatment for chronic abdominal pain.

However, there are some important critiques on this trial. First, a type II error by too low sample size cannot be excluded. Second, some experimental studies indicate that filmy adhesions, which may be disrupted by pneumoperitoneum in the control patient group, cause most pain. Third, adhesions might have reformed after adhesiolysis, diminishing long term effects in the adhesiolysis group. Adhesion formation and reformation can effectively be reduced by application of an anti-adhesion barrier. Apart from these critiques, there is no evidence for effective alternative treatments.

Patients with chronic postoperative pain are frequently referred to the outpatient clinical of the surgery department of the RadboudUMC for expert opinion. Since 2012 the investigators started a 'patient participation in care' project for this patient group, in which laparoscopic adhesiolysis was reintroduced as treatment for chronic abdominal in selected cases. Cine- MRI was used as a novel non-invasive tool to diagnose adhesions, waiving the need for a negative laparoscopy in patient with other causes for chronic abdominal pain. Cine- MRI was recently developed as a non-invasive diagnostic tool to detect symptomatic adhesions, with reported sensitivity between 85%- 89% and specificity between 93%-95%. Decision for operative treatment was made based on individualized assessment of benefits and risks based on cine-MRI results in a shared-decision approach. Further, all patients undergoing adhesiolysis were treated with an anti-adhesion barrier.

Purpose & Research question The aim of this study is to evaluate the results of this novel shared decision approach using cine-MRI in a cohort of patients referred to the outpatient clinical of the department of surgery with chronic postoperative pain. Comparison is made between patients undergoing laparoscopic adhesiolysis, patients conservatively treated with adhesions on cine-MRI, and patients with no adhesions on cine-MRI.

Patients: Patients with chronic postoperative pain (>6 months) caused by adhesions as proven by cine-MRI Intervention: Laparoscopic adhesiolysis with adhesion barrier Controls: - control group 1: Patients with chronic postoperative pain and cine-MRI proven adhesions who had conservative treatment - Control group 2 patients with alternative diagnosis who had conservative treatment Outcome: • Change in symptoms (measured by Patients' Global Impression of Change scale), current pain (measured by numeric rate scale), Healthcare utilization (hospital visits, paramedic visits, medication)

Plan of investigation We will perform an analysis in a cohort of approximately 100 patients who underwent Cine-MRI in the work-up for chronic abdominal pain. Adhesions were identified in approximately 80 of the patients, 40 of them were operated and underwent laparoscopic adhesiolysis (group 1). The other 40 patients waived operation for various reasons and received conservative treatment (group 2). Patients with negative cine-MRI are analyzed as group 3. In a few cases a diagnostic laparoscopy was performed in case history, physical examination and cine-MRI were inconclusive. These patients will be analyzed as part of group 1.

Patients will be asked to participate in this study by telephone or letter. If agreed, a questionnaire will be sent comparing pain, improvement of pain since treatment, use of analgesics and other healthcare utilization between the operated and non-operated groups. Further data on the operation and peri-operative complications are gathered from the case records. Primary outcome is reduction or alleviation of pain. Secondary outcomes are current pain score (measured by VAS), analgesics use and healthcare utilization. Additional secondary outcomes for the operatively treated group are the incidence of conversion to open surgery, and peri-operative complications.

Patients admitted to the outpatient clinic of the department of surgery for chronic postoperative pain who underwent a cine-MRI are screened for eligibility.

Inclusion criteria are :

* Age ≥ 18 years
* Pain exists for at least 6 months postoperatively

Exclusion criteria are:

- Cine-MRI not performed for chronic pain (e.g. recurrent pain with episodes of bowel obstructions)

ELIGIBILITY:
Inclusion criteria are :

* Age ≥ 18 years
* Pain exists for at least 6 months postoperatively

Exclusion criteria are:

- Cine-MRI not performed for chronic pain (e.g. recurrent pain with episodes of bowel obstructions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the outpatient clinic of the department of surgery for chronic postoperative pain who underwent a cine-MRI are screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in pain | long-term >6 months to 3 years following surgery or cineMRI
  measured by a verbal rating pain change scale (VRCS)

SECONDARY OUTCOMES:
Current pain | long-term >6 months to 3 years following surgery or cineMRI
  measured by visual analogue scale (VAS)
Frequency of pain | long-term >6 months to 3 years following surgery or cineMRI
  measured by a questionnaire using a seven-point Likert scale
Daily discomfort | long-term >6 months to 3 years following surgery or cineMRI
  measured by a questionnaire using a seven-point Likert scale
Healthcare utilization | long-term >6 months to 3 years following surgery or cineMRI
  measured by the number of visits to the general practitioner, medical specialist, paramedics and complementary practitioners
Complications of surgery/ adhesiolysis | Peri-operative (up to 30 days after adhesiolysis)
  registered and graded according to the Clavien-Dindo classification. Complications scored as Clavien-Dindo grade 3 or higher were considered severe complications.

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be made available for future research upon reasonable request

REFERENCES:
- [Background] ten Broek RP, Bakkum EA, Laarhoven CJ, van Goor H. Epidemiology and Prevention of Postsurgical Adhesions Revisited. Ann Surg. 2016 Jan;263(1):12-9. doi: 10.1097/SLA.0000000000001286. PMID 26135678
- [Background] Ten Broek RPG, Stommel MWJ, Strik C, van Laarhoven CJHM, Keus F, van Goor H. Benefits and harms of adhesion barriers for abdominal surgery: a systematic review and meta-analysis. Lancet. 2014 Jan 4;383(9911):48-59. doi: 10.1016/S0140-6736(13)61687-6. Epub 2013 Sep 27. PMID 24075279
- [Background] Gerner-Rasmussen J, Burcharth J, Gogenur I. The efficacy of adhesiolysis on chronic abdominal pain: a systematic review. Langenbecks Arch Surg. 2015 Jul;400(5):567-76. doi: 10.1007/s00423-015-1316-9. Epub 2015 Jun 20. PMID 26088873
- [Background] Swank DJ, Swank-Bordewijk SC, Hop WC, van Erp WF, Janssen IM, Bonjer HJ, Jeekel J. Laparoscopic adhesiolysis in patients with chronic abdominal pain: a blinded randomised controlled multi-centre trial. Lancet. 2003 Apr 12;361(9365):1247-51. doi: 10.1016/s0140-6736(03)12979-0. PMID 12699951
- [Background] Cheong YC, Reading I, Bailey S, Sadek K, Ledger W, Li TC. Should women with chronic pelvic pain have adhesiolysis? BMC Womens Health. 2014 Mar 4;14(1):36. doi: 10.1186/1472-6874-14-36. PMID 24588989
- [Result] van den Beukel BAW, Stommel MWJ, van Leuven S, Strik C, IJsseldijk MA, Joosten F, van Goor H, Ten Broek RPG. A Shared Decision Approach to Chronic Abdominal Pain Based on Cine-MRI: A Prospective Cohort Study. Am J Gastroenterol. 2018 Aug;113(8):1229-1237. doi: 10.1038/s41395-018-0158-9. Epub 2018 Jun 27. PMID 29946174
- Available data/document: Clinical Study Report — https://doi.org/10.1038/s41395-018-0158-9